CLINICAL TRIAL: NCT05141201
Title: Saphnelo for Intravenous Infusion 300 mg Specific Use Result Study All Patient Investigation in Patients With Systemic Lupus Erythematosus
Brief Title: SAPHNELO Systemic Lupus Erythematosus Japan Post-Marketing Surveillance (PMS)
Status: Active, not recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D3461C00022
Record Dates: First submitted 2021-11-19; First posted 2021-12-02 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Lupus Erythematosus, Systemic
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
To collect information on and evaluate the long-term safety and effectiveness of Anifrolumab in patients with systemic lupus erythematosus in the real-world post-marketing setting.

DETAILED DESCRIPTION:
The objective of the Specific Use Result Study is to collect information on and evaluate the long-term safety and effectiveness of Anifrolumab in patients with systemic lupus erythematosus insufficiently responding to currently available treatment in the real-world post-marketing setting.

This investigation will be conducted to support the application for re-examination specified in Article 14-4 of the Pharmaceutical Affairs Law.

ELIGIBILITY:
Inclusion Criteria:

patients with systemic lupus erythematosus insufficiently responding to currently available treatment -

Exclusion Criteria:

None

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with systemic lupus erythematosus insufficiently responding to currently available treatment
Sampling Method: Non-Probability Sample
Enrollment: 1620 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of ADRs | from the baseline to 52 weeks
  Incidence of ADRs related to Anifrolimab. Safety specification: Herpes zoster, serious infections, anaphylaxis, malignancy and reactivation of hepatitis B virus

CONTACTS AND LOCATIONS:
Locations (47):
- Japan (47):
  - Research Site, Aichi
  - Research Site, Akita
  - Research Site, Aomori
  - Research Site, Chiba
  - Research Site, Ehime
  - Research Site, Fukui
  - Research Site, Fukuoka
  - Research Site, Fukushima
  - Research Site, Gifu
  - Research Site, Gunma
  - Research Site, Hiroshima
  - Research Site, Hokkaido
  - Research Site, Hyōgo
  - Research Site, Ibaraki
  - Research Site, Ishikawa
  - Research Site, Kagawa
  - Research Site, Kagoshima
  - Research Site, Kanagawa
  - Research Site, Kochi
  - Research Site, Kumamoto
  - Research Site, Kyoto
  - Research Site, Mie
  - Research Site, Miyagi
  - Research Site, Miyazaki
  - Research Site, Nagano
  - Research Site, Nagasaki
  - Research Site, Nara
  - Research Site, Niigata
  - Research Site, Numakunai
  - Research Site, Okayama
  - Research Site, Okinawa
  - Research Site, Osaka
  - Research Site, Ōita
  - Research Site, Saga
  - Research Site, Saitama
  - Research Site, Shiga
  - Research Site, Shimane
  - Research Site, Shizuoka
  - Research Site, Tochigi
  - Research Site, Tokushima
  - Research Site, Tokyo
  - Research Site, Tottori
  - Research Site, Toyama
  - Research Site, Wakayama
  - Research Site, Yamagata
  - Research Site, Yamaguchi
  - Research Site, Yamanashi

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluatedas per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes,indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level datain an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access.For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home